CLINICAL TRIAL: NCT03696160
Title: An Open-Label, Multi-Centre, Randomised Study to Investigate Integrase Inhibitor Versus Boosted Protease Inhibitor Antiretroviral Therapy for Patients With Advanced HIV Disease
Brief Title: The Late Presenter Treatment Optimisation Study
Acronym: LAPTOP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: NEAT ID Foundation (Other)
Collaborators: Gilead Sciences (Industry); Janssen Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NEAT44
Record Dates: First submitted 2018-09-24; First posted 2018-10-04 (Actual); Results first posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: HIV/AIDS
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — bictegravir, emtricitabine, tenofovir alafenamide, drug combination; symtuza

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Biktarvy (Experimental): Bictegravir is an inhibitor of HIV-1 integrase that is being evaluated for the treatment of HIV-1 infection.
  Biktarvy® received marketing authorisation valid throughout the European Union (EU) in June 2018.
  Biktarvy is a combination of bictegravir, emtricitabine, and tenofovir (B/F/TAF).
  Method of administration: One combined B 50mg/F 200mg/TAF 25mg tablet taken orally once daily for up to 48 weeks without regard to food.
  Interventions: Drug: Biktarvy
- Symtuza (Experimental): Symtuza® is a boosted PI indicated for the treatment of HIV-1 infection.
  Symtuza® received marketing authorisation valid throughout the EU in September 2017.
  Symtuza is a combination of darunavir, cobicistat, emtricitabine and tenofovir alafenamide (D/C/F/TAF)
  Method of administration: One combined D 800mg/C 150mg/F 200mg/TAF 10mg tablet taken orally once daily for up to 48 weeks with the addition of food.
  Interventions: Drug: Symtuza

INTERVENTIONS:
Drug: Biktarvy — Integrase inhibitor used to treat HIV-1 infection
  Arms: Biktarvy
Drug: Symtuza — Protease inhibitor used to treat HIV-1 infection
  Arms: Symtuza

SUMMARY:
The main purpose of this study is to compare two different types of HIV treatments, in terms of effectiveness and improvement of side effects, for patients who are diagnosed with a more advanced HIV infection. Patients with advanced HIV infections are otherwise known as 'late presenters'.

There are many effective treatments for HIV available; however, for late presenting patients the investigators do not know which type of treatment performs best. This is the first large study to compare treatments for patients in this situation, and the investigators hope that the results of this study will help doctors decide which treatments to use in the future.

The two different types of treatment the investigators are comparing both contain a mixture of drugs that work together to combat HIV:

The Boosted Protease Inhibitor combination (PI) which is a combination tablet containing: darunavir, cobicistat, emtricitabine and tenofovir alafenamide. It was approved for use in Europe under the brand name Symtuza®.

The Integrase Inhibitor combination (INI). Which is a combination tablet containing: bictegravir, emtricitabine and tenofovir alafenamide. This is a a newer combination which was approved for use in Europe in June 2018 under the brand name of Biktarvy®.

The main difference between the two treatments is how each one fights a HIV infection. They both stop a part of the virus from working (i.e. inhibit it), to prevent it from making copies of itself. The PI treatment contains drugs to stop the protease part of the virus, whereas the INI treatment contains drugs to stop the integrase part.

In recent studies, it appears that treatments containing integrase inhibitors may be better for late presenting patients. They have been shown to quickly bring down the amount of virus in the body, and the side effects may be more acceptable to late presenters.

To compare the two treatments, half of the participants on this study will be given the PI treatment, and the other half will be given the INI treatment.

DETAILED DESCRIPTION:
The effectiveness of HIV antiretroviral therapy (ART) has consistently improved over the years. This is largely due to newer drugs having improved antiviral effectiveness and more tolerable side effect profiles; resulting in better viral suppression and improved treatment adherence. On the other hand, most recent clinical trials look at the effectiveness of ART in patients with less advanced disease. These patients usually suffer from less related diseases, drug-drug interactions, and other risks for treatment failure. Outside of these trials, the number of patients who present to clinic with a more developed advanced HIV infection, known as 'late presenters', remains high across Europe. Trials for these patients have tended to focus on the time of starting treatment and the management of infections.

Much less is known about which ART treatments perform best for these late presenting patients; particularly in terms of virus suppression, immune system recovery, side effects and improvement of AIDs related diseases. No specific drug combinations have been compared in appropriate clinical trials before, and the international guidelines for first line treatment judge all therapies as equal standard of care for these patients.

The investigators anticipate that Integrase inhibitor containing regimes may be better suited to patients with advanced disease, due to their beneficial side-effect profile and ability to rapidly decrease viral load levels. Therefore the investigators are conducting this clinical trial to compare an integrase inhibitor regime, against a protease inhibitor regime in patients with advanced HIV infection. The aim of the study is to demonstrate the non-inferiority of Biktarvy® against Symtuza®.

Patients will be recruited from sites across Europe, and randomized onto either arm of the study. After randomisation onto either treatment regime, patients will attend approximately 9 follow-up visits over the course of a year. During these visits, patients will be asked to complete two questionnaires, to assess their quality of life and HIV symptoms. They will also be asked to provide a number of blood samples. These samples are to ensure that the patient is not resistant to the study drug and that their disease is not worsening. Samples to test for study drug resistance will be shipped to a laboratory for analysis in the even that the patient experiences virological failure.

Biktarvy® will be supplied from Gilead and Symtuza® will be provided by Janssen Pharmaceuticals.

ELIGIBILITY:
Inclusion Criteria:

1. The ability to understand and sign a written informed consent form (ICF) and must be willing to comply with all study requirements.
2. Male or non-pregnant, non-lactating females†.
3. Age ≥ 18 years.
4. Have documented, untreated HIV-1 infection with either:

   1. AIDS with any CD4 cell count (AIDS-defining conditions are listed within Appendix 3).

      Or
   2. Severe bacterial infection (BI)‡ and must have a CD4 cell count < 200/μl within 28 days prior to study entry§.

      Or
   3. Any symptoms or no symptoms and must have a CD4 cell count < 100/μL within 28 days prior to study entry and must have an entry HIV viral load > 1000 copies/mL.

      Or
   4. Currently receiving treatment for OI**. i. Subjects with other serious OIs, including other AIDS-defining and AIDS-related OIs for which appropriate therapy other than ART exists are eligible, but Investigator approval must be obtained. ii. Current OI treatment can have been discontinued prior to start of ART.
5. Have an entry HIV viral load > 1000 copies/mL
6. Have the ability to take oral medications.
7. Females of childbearing potential and heterosexually active males must be willing to use a highly effective method of contraception and be willing to continue practising these birth control methods during the trial and for at least 30 days after the last dose of study medication. See Appendix 7 for further details.

Such methods include:

* True abstinence from penile-vaginal intercourse, when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods), and withdrawal are not acceptable methods of contraception).
* Non-hormonal Intrauterine device or non-hormonal intrauterine system that meets the effectiveness criteria as stated in the product label.
* Male partner sterilization prior to the female subject's entry into the study, and this male is the sole partner for that subject.
* Combined (oestrogen and progesterone containing) hormonal contraception associated with the inhibition of ovulation*:
* Oral
* Intravaginal
* Transdermal
* Bilateral tubal occlusion

Exclusion Criteria:

1. Any therapeutic ARV which commenced less than 2 weeks prior to screening and which was taken for more than 48 hours
2. Systemic cancer chemotherapy within 30 days prior to study entry, or current treatment for cancer (with the exception of Kaposi's sarcoma) or lymphoma.
3. Current or anticipated use of contraindicated medications (see Summary of Product Characteristics (SmPC) for Symtuza® and Biktarvy®) or anticipated systemic chemotherapy during study enrolment (administration of any contraindicated medication must be discontinued at least 30 days prior to the baseline visit and for the duration of the study).
4. Known resistance to the components of study medications (see section 6.1.3 for more details).
5. History or symptoms of advanced renal and/or hepatic impairment. Such as, kidney failure requiring dialysis; eGFR <30 mL/min; hepatic transaminases (AST and ALT) > 5 x upper limit of normal (ULN); or, platelet count <50,000.
6. Current drug or alcohol use that, in the opinion of the Investigator, would cause interference with the study.
7. Cryptococcal meningitis or active TB, or current or expected treatment requiring Rifampicin or Rifabutin (patients with expected latent TB will have a TB test (IGRAs e.g. ELISPOT, QuantiFERON etc.) at their screening visit).
8. History or presence of allergy to the study drugs or their components, or drugs of their class.
9. Using any concomitant therapy disallowed as per the product labelling for the study drugs.
10. Any investigational drug within 30 days prior to the study drug administration.
11. Patients with severe (Child Pugh class C) hepatic impairment.
12. Women who are pregnant, breastfeeding or plan to become pregnant or breastfeed during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 447 (Actual)
Dates: Start 2019-03-05 (Actual); Primary Completion 2024-06-17 (Actual); Study Completion 2024-06-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Georg Behrens, Study Director — Hannover Medical School
Locations (53):
- Belgium (3):
  - Institute of Tropical Medicine, Antwerp
  - CHU Saint-Pierre, Brussels
  - University Hospital Ghent, Ghent
- France (8):
  - Hopital Europeen Marseille, Marseille
  - Groupe Hospitalier Sud Ile-de-France (Melun), Melun
  - Hôpital Gui de Chauliac, Montpellier
  - CHU de Nantes, Nantes
  - Hopital Lariboisiere, Paris
  - Hopital Saint-Louis, Paris
  - Hôpital Saint Antoine, Paris
  - Pitié-Salpêtrière Hospital, Paris
- Germany (7):
  - Medizinische Klinik und Poliklinik Universitätsklinikum Bonn, Bonn
  - University Hospital Koln, Cologne
  - Goethe University Hospital Frankfurt, Frankfurt
  - University Hospital Geissen, Geißen
  - ICH Study Center Gmbh & Co. KG, Hamburg
  - Medizinische Hochschule Hannover, Hanover
  - University Hospital Klinikum rechts der Isar der TUM, Munich
- Ireland (2):
  - Mater Misericordiae University Hospital, Dublin
  - St Vincent's University Hospital, Dublin
- Italy (5):
  - Luigi Sacco Hospital, Milan
  - Ospedale San Raffaele, Milan
  - ASST Santi Paolo, Milan
  - Clinica of Infectious Diseases, Modena
  - INMI Lazzaro Spallanzani, Rome, Rome
- Spain (13):
  - Hospital General Universatario Alicante, Alicante
  - Hospital Bellvitge, Barcelona
  - Hospital Clinic (Helios Building), Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital del Mar, Barcelona
  - Hospital Trias i Pujol, Barcelona
  - Hospital Universitari Vall d'Herbon, Barcelona
  - Hospital General Universitatrio de Elche, Elche
  - Hospital 12 Octubre, Madrid
  - Hospital de la Princesa, Madrid
  - Hospital Ramon y Cajal, Madrid
  - Hospital Universitatrio La Paz, Madrid
  - Hospital Virgen de la Victoria, Málaga
- United Kingdom (15):
  - Royal Bournemouth Hospital, Bournemouth
  - Southmead Hospital, Bristol
  - Leeds Teaching Hospital, Leeds
  - Barts Health, London
  - Chelsea and Westminister, London
  - Guy's Hospital, London
  - Homerton University Hospital, London
  - Imperial College Healthcare Trust, London
  - Kings College London, London
  - Mortimer Market Centre, London
  - Royal Free Hospital, London
  - St George's Hospital, London
  - University Hospital Lewisham, London
  - North Manchester General Hospital, Manchester
  - Sheffield Teaching Hospital, Sheffield

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] DeJesus E, Rockstroh JK, Henry K, Molina JM, Gathe J, Ramanathan S, Wei X, Yale K, Szwarcberg J, White K, Cheng AK, Kearney BP; GS-236-0103 Study Team. Co-formulated elvitegravir, cobicistat, emtricitabine, and tenofovir disoproxil fumarate versus ritonavir-boosted atazanavir plus co-formulated emtricitabine and tenofovir disoproxil fumarate for initial treatment of HIV-1 infection: a randomised, double-blind, phase 3, non-inferiority trial. Lancet. 2012 Jun 30;379(9835):2429-2438. doi: 10.1016/S0140-6736(12)60918-0. PMID 22748590
- [Background] Raffi F, Rachlis A, Stellbrink HJ, Hardy WD, Torti C, Orkin C, Bloch M, Podzamczer D, Pokrovsky V, Pulido F, Almond S, Margolis D, Brennan C, Min S; SPRING-2 Study Group. Once-daily dolutegravir versus raltegravir in antiretroviral-naive adults with HIV-1 infection: 48 week results from the randomised, double-blind, non-inferiority SPRING-2 study. Lancet. 2013 Mar 2;381(9868):735-43. doi: 10.1016/S0140-6736(12)61853-4. Epub 2013 Jan 8. PMID 23306000
- [Background] Walmsley SL, Antela A, Clumeck N, Duiculescu D, Eberhard A, Gutierrez F, Hocqueloux L, Maggiolo F, Sandkovsky U, Granier C, Pappa K, Wynne B, Min S, Nichols G; SINGLE Investigators. Dolutegravir plus abacavir-lamivudine for the treatment of HIV-1 infection. N Engl J Med. 2013 Nov 7;369(19):1807-18. doi: 10.1056/NEJMoa1215541. PMID 24195548
- [Background] Sax et al. Phase 3 Randomized, Controlled, Clinical Trial of Bictegravir Coformulated With FTC/TAF in a Fixed-Dose Combination vs Dolutegravir + FTC/TAF in Treatment-Naïve HIV-1-Positive Adults: Week 48 Results. 9th IAS Conference on HIV Science; Paris, France; July 23-26, 2017
- [Background] Gallant et al. A phase 3 randomized controlled clinical trial of bictegravir in a fixed dose combination, B/F/TAF, vs ABC/DTG/3TC in treatment-naïve adults at week 48. 9th IAS Conference on HIV Science; Paris, France; July 23-26, 2017. MOAB0105LB
- [Background] Camoni L, Raimondo M, Regine V, Salfa MC, Suligoi B; regional representatives of the HIV Surveillance System. Late presenters among persons with a new HIV diagnosis in Italy, 2010-2011. BMC Public Health. 2013 Mar 27;13:281. doi: 10.1186/1471-2458-13-281. PMID 23537210
- [Background] Montlahuc C, Guiguet M, Abgrall S, Daneluzzi V, de Salvador F, Launay O, Martinez V, Partisani M, Pradier C, Rouveix E, Valin N, Grabar S, Costagliola D; French Hospital Database ANRS CO4 cohort. Impact of late presentation on the risk of death among HIV-infected people in France (2003-2009). J Acquir Immune Defic Syndr. 2013 Oct 1;64(2):197-203. doi: 10.1097/QAI.0b013e31829cfbfa. PMID 24047970
- [Background] Antinori A, Coenen T, Costagiola D, Dedes N, Ellefson M, Gatell J, Girardi E, Johnson M, Kirk O, Lundgren J, Mocroft A, D'Arminio Monforte A, Phillips A, Raben D, Rockstroh JK, Sabin C, Sonnerborg A, De Wolf F; European Late Presenter Consensus Working Group. Late presentation of HIV infection: a consensus definition. HIV Med. 2011 Jan;12(1):61-4. doi: 10.1111/j.1468-1293.2010.00857.x. PMID 20561080
- [Background] Raffetti E, Postorino MC, Castelli F, Casari S, Castelnuovo F, Maggiolo F, Di Filippo E, D'Avino A, Gori A, Ladisa N, Di Pietro M, Sighinolfi L, Zacchi F, Torti C. The risk of late or advanced presentation of HIV infected patients is still high, associated factors evolve but impact on overall mortality is vanishing over calendar years: results from the Italian MASTER Cohort. BMC Public Health. 2016 Aug 25;16(1):878. doi: 10.1186/s12889-016-3477-z. PMID 27557878
- [Background] Sobrino-Vegas P, Rodriguez-Urrego J, Berenguer J, Caro-Murillo AM, Blanco JR, Viciana P, Moreno S, Bernardino I, del Amo J; CoRIS. Educational gradient in HIV diagnosis delay, mortality, antiretroviral treatment initiation and response in a country with universal health care. Antivir Ther. 2012;17(1):1-8. doi: 10.3851/IMP1939. PMID 22267463
- [Background] Late presenters working group in COHERE in EuroCoord; Mocroft A, Lundgren J, Antinori A, Monforte Ad, Brannstrom J, Bonnet F, Brockmeyer N, Casabona J, Castagna A, Costagliola D, De Wit S, Fatkenheuer G, Furrer H, Jadand C, Johnson A, Lazanas M, Leport C, Moreno S, Mussini C, Obel N, Post F, Reiss P, Sabin C, Skaletz-Rorowski A, Suarez-Loano I, Torti C, Warszawski J, Wittkop L, Zangerle R, Chene G, Raben D, Kirk O. Late presentation for HIV care across Europe: update from the Collaboration of Observational HIV Epidemiological Research Europe (COHERE) study, 2010 to 2013. Euro Surveill. 2015;20(47). doi: 10.2807/1560-7917.ES.2015.20.47.30070. PMID 26624933
- [Background] Abdool Karim SS, Naidoo K, Grobler A, Padayatchi N, Baxter C, Gray AL, Gengiah T, Gengiah S, Naidoo A, Jithoo N, Nair G, El-Sadr WM, Friedland G, Abdool Karim Q. Integration of antiretroviral therapy with tuberculosis treatment. N Engl J Med. 2011 Oct 20;365(16):1492-501. doi: 10.1056/NEJMoa1014181. PMID 22010915
- [Background] Blanc FX, Sok T, Laureillard D, Borand L, Rekacewicz C, Nerrienet E, Madec Y, Marcy O, Chan S, Prak N, Kim C, Lak KK, Hak C, Dim B, Sin CI, Sun S, Guillard B, Sar B, Vong S, Fernandez M, Fox L, Delfraissy JF, Goldfeld AE; CAMELIA (ANRS 1295-CIPRA KH001) Study Team. Earlier versus later start of antiretroviral therapy in HIV-infected adults with tuberculosis. N Engl J Med. 2011 Oct 20;365(16):1471-81. doi: 10.1056/NEJMoa1013911. PMID 22010913
- [Background] Zolopa A, Andersen J, Powderly W, Sanchez A, Sanne I, Suckow C, Hogg E, Komarow L. Early antiretroviral therapy reduces AIDS progression/death in individuals with acute opportunistic infections: a multicenter randomized strategy trial. PLoS One. 2009;4(5):e5575. doi: 10.1371/journal.pone.0005575. Epub 2009 May 18. PMID 19440326
- [Background] Mussini C, Manzardo C, Johnson M, Monforte Ad, Uberti-Foppa C, Antinori A, Gill MJ, Sighinolfi L, Borghi V, Lazzarin A, Miro JM, Sabin C; Late Presenter Investigators. Patients presenting with AIDS in the HAART era: a collaborative cohort analysis. AIDS. 2008 Nov 30;22(18):2461-9. doi: 10.1097/QAD.0b013e328314b5f1. PMID 19005269
- [Background] Demarest J, Underwood M, St Clair M, Dorey D, Brown D, Zolopa A. Short Communication: Dolutegravir-Based Regimens Are Active in Integrase Strand Transfer Inhibitor-Naive Patients with Nucleoside Reverse Transcriptase Inhibitor Resistance. AIDS Res Hum Retroviruses. 2018 Apr;34(4):343-346. doi: 10.1089/AID.2017.0184. Epub 2018 Mar 22. PMID 29444582
- [Background] Wijting I et al. Integrase Inhibitors are an Independent Risk Factor for IRIS: An ATHENA Cohort Study. Conference on Retroviruses and Opportunistic Infections. February 2017. Seattle, WA, USA. Abstract 731.
- [Background] Dutertre M et al. Initiation of ART Based on Integrase Inhibitors Increases the Risk of IRIS. Conference on Retroviruses and Opportunistic Infections. February 2017. Seattle, WA, USA. Abstract 732.
- [Background] Psichogiou M, Basoulis D, Tsikala-Vafea M, Vlachos S, Kapelios CJ, Daikos GL. Integrase Strand Transfer Inhibitors and the Emergence of Immune Reconstitution Inflammatory Syndrome (IRIS). Curr HIV Res. 2017;15(6):405-410. doi: 10.2174/1570162X15666171122155708. PMID 29173177
- [Background] Hill AM, Mitchell N, Hughes S, Pozniak AL. Risks of cardiovascular or central nervous system adverse events and immune reconstitution inflammatory syndrome, for dolutegravir versus other antiretrovirals: meta-analysis of randomized trials. Curr Opin HIV AIDS. 2018 Mar;13(2):102-111. doi: 10.1097/COH.0000000000000445. PMID 29278532
- [Background] Paredes R, Tzou PL, van Zyl G, Barrow G, Camacho R, Carmona S, Grant PM, Gupta RK, Hamers RL, Harrigan PR, Jordan MR, Kantor R, Katzenstein DA, Kuritzkes DR, Maldarelli F, Otelea D, Wallis CL, Schapiro JM, Shafer RW. Collaborative update of a rule-based expert system for HIV-1 genotypic resistance test interpretation. PLoS One. 2017 Jul 28;12(7):e0181357. doi: 10.1371/journal.pone.0181357. eCollection 2017. PMID 28753637
- [Background] Levy et al. ANRS 146 - GeSIDA 7211 OPTIMAL phase III trial: maraviroc plus cART in advanced HIV-1-infected individuals. Journal Of The International Aids Society (Vol. 20, Pp. 6-7)
- [Background] Slama L, Landman R, Assoumou L, Benalycherif A, Samri A, Joly V, Pialoux G, Valin N, Cabie A, Duvivier C, Lambert-Niclot S, Marcelin AG, Peytavin G, Costagliola D, Girard PM; IMEA 040 DATA Study Group. Efficacy and safety of once-daily ritonavir-boosted atazanavir or darunavir in combination with a dual nucleos(t)ide analogue backbone in HIV-1-infected combined ART (cART)-naive patients with severe immunosuppression: a 48 week, non-comparative, randomized, multicentre trial (IMEA 040 DATA trial). J Antimicrob Chemother. 2016 Aug;71(8):2252-61. doi: 10.1093/jac/dkw103. Epub 2016 Apr 10. PMID 27068399
- [Derived] Behrens GMN, Assoumou L, Liegeon G, Antinori A, Mican R, Genderini FG, Post FA, Rockstroh JK, Hamzah L, Domingo P, Curran A, Laguno M, Fletcher C, Moody J, Pozniak A; NEAT-ID Foundation; LAPTOP Study Team. Integrase versus protease inhibitor therapy in advanced HIV disease (LAPTOP): a multicountry, randomised, open-label, non-inferiority trial. Lancet Infect Dis. 2025 Dec 1:S1473-3099(25)00681-4. doi: 10.1016/S1473-3099(25)00681-4. Online ahead of print. PMID 41344354

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Number of Subjects Enrolled: 447
Pre-assignment Details: Number of Subjects Screened: 475
Period: Overall Study
Arm/Group | Biktarvy | Symtuza
Started | 222 | 225
Completed | 220 | 222
Not Completed | 2 | 3
Not completed — Withdrew before IMP dosing | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Biktarvy | Symtuza | Total
Number analyzed (Participants) | 220 | 222 | 442
Age, Continuous [Median (Inter-Quartile Range); unit: Years] — >18 years
  Years | 44 [36 to 54] | 42 [34 to 51] | 43 [35 to 53]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 44 | 84
  Male | 180 | 178 | 358
Region of Enrollment [Number; unit: Participants]
  United Kingdom | 45 | 42 | 87
  Spain | 61 | 61 | 122
  France | 30 | 32 | 62
  Belgium | 17 | 17 | 34
  Italy | 28 | 30 | 58
  Germany | 37 | 38 | 75
  Ireland | 2 | 2 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants] — White, Black, Other
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 43 | 40 | 83
    White | 140 | 136 | 276
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 37 | 46 | 83

OUTCOME MEASURES:

1. Primary Outcome: Treatment Failure
Description: Composite outcome: treatment failure due to either virological or clinical reasons. Virological reasons can either be insufficient virological response or viral rebound. Clinical reasons can be death related to HIV/AIDS/opportunistic infection or severe bacterial infection, new or recurrent AIDS defining event, any serious non-AIDS defining event or clinically relevant adverse events of any grade or immune reconstitution inflammatory syndrome requiring treatment
Time Frame: Earliest at 12 weeks, latest 48 weeks
Population: Each row represents a different analysis using different patient numbers, dependent on mITT or PP analysis
Measure: Count of Participants; unit: Participants
Groups:
- Biktarvy: Bictegravir is an inhibitor of HIV-1 integrase that is being evaluated for the treatment of HIV-1 infection.
  Biktarvy® received marketing authorisation valid throughout the European Union (EU) in June 2018.
  Biktarvy is a combination of bictegravir, emtricitabine, and tenofovir (B/F/TAF).
  Method of administration: One combined B 50mg/F 200mg/TAF 25mg tablet taken orally once daily for up to 48 weeks without regard to food.
  Biktarvy: Integrase inhibitor used to treat HIV-1 infection
- Symtuza: Symtuza® is a boosted PI indicated for the treatment of HIV-1 infection.
  Symtuza® received marketing authorisation valid throughout the EU in September 2017.
  Symtuza is a combination of darunavir, cobicistat, emtricitabine and tenofovir alafenamide (D/C/F/TAF)
  Method of administration: One combined D 800mg/C 150mg/F 200mg/TAF 10mg tablet taken orally once daily for up to 48 weeks with the addition of food.
  Symtuza: Protease inhibitor used to treat HIV-1 infection
Arm/Group | Biktarvy | Symtuza
Number analyzed (Participants) | 220 | 222
Participants
  mITT analysis | 49 | 70
  PP analysis: number analyzed (Participants) | 219 | 222
  PP analysis | 48 | 69

2. Secondary Outcome: Proportion of Patients With HIV-RNA Viral Load <50 Copies/mL
Description: at week 24, 36, 48
Time Frame: Week 24, 36 and 48
Measure: Count of Participants; unit: Participants
Arm/Group | Biktarvy | Symtuza
Number analyzed (Participants) | 220 | 222
Participants
  <50 at Week 24 | 127 | 112
  <50 at Week 36 | 135 | 134
  <50 at Week 48 | 151 | 136

3. Secondary Outcome: Time to Reach CD4 (Cluster of Differentiation 4) Count >200/µL
Time Frame: Through study completion, up to 48 weeks.
Measure: Count of Participants; unit: Participants
Arm/Group | Biktarvy | Symtuza
Number analyzed (Participants) | 220 | 222
Participants
  CD4 >200 W0 | 9 | 8
  CD4 >200 W4 | 65 | 58
  CD4 >200 W8 | 72 | 65
  CD4 >200 W12 | 74 | 71
  CD4 >200 W24 | 87 | 91
  CD4 >200 W36 | 110 | 114
  CD4 >200 W48 | 115 | 121

4. Secondary Outcome: Proportion of Patients With CD4 Cell Count <200 and < 350μL at Week 4, 8, 12, 24, 36, 48
Time Frame: 4, 8, 12, 24, 36, 48 weeks
Population: Number analysed differs due to:
  * some CD4 tests missed at visit
  * some patients withdraw/miss visits
Measure: Count of Participants; unit: Participants
Arm/Group | Biktarvy | Symtuza
Number analyzed (Participants) | 220 | 222
Participants
  <200 at W4: number analyzed (Participants) | 201 | 211
  <200 at W4 | 136 | 153
  <200 at W8: number analyzed (Participants) | 186 | 201
  <200 at W8 | 114 | 136
  <200 at W12: number analyzed (Participants) | 190 | 204
  <200 at W12 | 116 | 133
  <200 at W24: number analyzed (Participants) | 188 | 198
  <200 at W24 | 101 | 107
  <200 at W36: number analyzed (Participants) | 186 | 195
  <200 at W36 | 76 | 81
  <200 at W48: number analyzed (Participants) | 179 | 186
  <200 at W48 | 64 | 65
  <350 at W4: number analyzed (Participants) | 201 | 211
  <350 at W4 | 185 | 195
  <350 at W8: number analyzed (Participants) | 186 | 201
  <350 at W8 | 162 | 187
  <350 at W12: number analyzed (Participants) | 190 | 204
  <350 at W12 | 165 | 190
  <350 at W24: number analyzed (Participants) | 188 | 198
  <350 at W24 | 160 | 180
  <350 at W36: number analyzed (Participants) | 186 | 195
  <350 at W36 | 152 | 161
  <350 at W48: number analyzed (Participants) | 179 | 186
  <350 at W48 | 137 | 151

5. Secondary Outcome: CD4/CD8 (Cluster of Differentiation 8) Ratio
Description: CD4/CD8 ratio at week 4, 8, 12, 24, 36, 48
Time Frame: Week 4, 8, 12, 24, 36, 48
Population: Number analysed differs due to:
  * some CD4:CD8 tests missed at visit
  * some patients withdraw/miss visits
Measure: Mean (Standard Error); unit: Ratio
Arm/Group | Biktarvy | Symtuza
Number analyzed (Participants) | 220 | 222
Ratio
  Week 0: number analyzed (Participants) | 216 | 222
  Week 0 | 0.11 (0.01) | 0.11 (0.01)
  Week 4: number analyzed (Participants) | 196 | 209
  Week 4 | 0.2 (0.01) | 0.18 (0.01)
  Week 8: number analyzed (Participants) | 182 | 200
  Week 8 | 0.2 (0.01) | 0.19 (0.01)
  Week 12: number analyzed (Participants) | 189 | 203
  Week 12 | 0.22 (0.01) | 0.2 (0.01)
  Week 24: number analyzed (Participants) | 185 | 196
  Week 24 | 0.27 (0.01) | 0.25 (0.01)
  Week 36: number analyzed (Participants) | 182 | 193
  Week 36 | 0.31 (0.01) | 0.28 (0.01)
  Week 48: number analyzed (Participants) | 179 | 184
  Week 48 | 0.33 (0.01) | 0.31 (0.01)

6. Secondary Outcome: Incidence of Immune Reconstitution Inflammatory Syndrome
Description: Incidence of Immune Reconstitution Inflammatory Syndrome
Time Frame: Week 48
Measure: Count of Participants; unit: Participants
Arm/Group | Biktarvy | Symtuza
Number analyzed (Participants) | 220 | 222
Participants | 7 | 8

7. Secondary Outcome: Number of Participants With Hospitalisation or Relapse of Specific Opportunistic or Bacterial Infection
Description: Start/Stop of hospitalization for any reason Start/Stop of opportunistic infections as listed within Appendix 3 (AIDS defining events according to https://www.cdc.gov/mmwr/preview/mmwrhtml/rr5710a2.htm) Start/Stop of severe BI, which consists of any of bacterial pneumonia, invasive bacterial infection (IBI) or any bacterial infectious disorder with grade 3 severity or requiring unscheduled hospital admission. An IBI is defined as the isolation of a bacterial organism from a normally sterile body site, or for bacterial nucleic acid to be detected at a normally sterile body site. Sterile body sites include blood, cerebrospinal fluid, pleural fluid, pericardial fluid, peritoneal fluid, joint fluid, bone aspirate, or a deep tissue abscess.
Time Frame: Week 48
Measure: Count of Participants; unit: Participants
Arm/Group | Biktarvy | Symtuza
Number analyzed (Participants) | 220 | 222
Participants | 41 | 53

8. Secondary Outcome: Number of Participants With Treatment-related Adverse Events as Assessed by Division of AIDS Adverse Event (AE) Grading Table Corrected Version 2.1-July 2017
Time Frame: Week 48
Measure: Count of Participants; unit: Participants
Arm/Group | Biktarvy | Symtuza
Number analyzed (Participants) | 220 | 222
Participants
  Any AE's ≥Grade 2 | 124 | 139
  Grade 2 AE's | 111 | 127
  Grade 3 AE's | 37 | 46
  Grade 4 AE's | 18 | 13
  Grade 3 or 4 AE's | 47 | 52
  Drug-Related AE's ≥Grade 2 | 16 | 32
  Drug-Related AE's Grade 3 or 4 | 3 | 4
  AE's leading to study drug interruption | 16 | 18
  SAE's | 48 | 52
  Death | 9 | 3

9. Secondary Outcome: ART and OI/BI Treatment Changes and Dose Modifications Due to Toxicities and DDI With ART, and IRIS Through Week 48
Description: Antiretroviral therapy and opportunistic or bacterial infection treatment changes and dose modifications due to toxicities and drug-drug interaction with antiretroviral therapy, and Immune Reconstitution Inflammatory Syndrome
Time Frame: Week 48
Measure: Count of Participants; unit: Participants
Arm/Group | Biktarvy | Symtuza
Number analyzed (Participants) | 220 | 222
Participants
  % of participants with ART change or study discontinuation due to toxicities, DDI, or IRIS | 23 | 19
  ART change or study discontinuation due to toxicities | 11 | 12
  ART change or study discontinuation due to IRIS | 2 | 1
  ART change or study discontinuation due to DDI | 10 | 6

10. Secondary Outcome: Health Care Resource Use, Including Number of Participants With Critical Care and Emergency Room Visits
Time Frame: Week 48
Measure: Count of Participants; unit: Participants
Arm/Group | Biktarvy | Symtuza
Number analyzed (Participants) | 220 | 222
Participants
  Incidence of critical care admission | 3 | 2
  Incidence of emergency room | 28 | 33

11. Secondary Outcome: QOL and Functional Status Outcomes, Including Overall Self-reported QOL and Functional Status Compared in the Two Groups at Week 48
Description: EQ-5D-3L (European Quality of life - 5 Dimensions - 3 Levels) and HIV Symptoms Index questionnaires will be completed by patients throughout the study to assess any change throughout their treatment
  Quality of life (EQ-5D-3L questionnaire) Scale is VAS Score which runs from 0 (worst health imaginable) to 100 (best health imaginable). We report the mean change from Baseline to W48.
  The HIV Symptom Index score is the sum of frequency ratings for the 20 selected symptoms; the score could range from 0 to 80 (80 being worst score). We report the mean change from Baseline to W48.
Time Frame: Week 48
Measure: Mean (Standard Error); unit: Questionnaire Score
Arm/Group | Biktarvy | Symtuza
Number analyzed (Participants) | 220 | 222
Questionnaire Score
  Quality of life (EQ-5D-3L questionnaire) Mean difference from Baseline to W48 | 20.6 (1.5) | 16.9 (1.5)
  HIV Symptoms Index Mean difference from Baseline to W48 | -12.0 (0.9) | -9.9 (0.8)

12. Secondary Outcome: Discontinuation or Modification of Study Medication Due to Insufficient Virological Response or Resistance Mutation Development
Description: Discontinuation or modification of the single tablet regimen due virological reasons defined as a) Insufficient virological response, either:
  1. HIV-1 RNA reduction < 1 log 10 copies/mL at week 12, or
  2. Viral load > 50 HIV-1 RNA copies/mL at week 48 b) Viral rebound, which is subsequently confirmed at the following scheduled or unscheduled visit, defined as either:
  a. Rebound of HIV-1 RNA to >200 copies/mL after having achieved HIV-1 RNA <50 copies/mL b. Rebound of HIV RNA by >1 log 10 copies/mL from nadir value, for patients whose viral load has never been suppressed below 50 copies/mL
Time Frame: Week 48
Measure: Count of Participants; unit: Participants
Arm/Group | Biktarvy | Symtuza
Number analyzed (Participants) | 220 | 222
Participants
  Participants with ART change or discontinuation due to virological response or resistance mutations | 3 | 1
  ART change or study discontinuation due to resistance mutations | 2 | 1
  ART change or study discontinuation due to insufficient virological response | 1 | 0

13. Secondary Outcome: Duration of Hospitalisations
Description: Duration of hospitalization for any reason
Time Frame: Week 48
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Biktarvy | Symtuza
Number analyzed (Participants) | 220 | 222
Days | 10 [6 to 14] | 13 [10 to 16]

ADVERSE EVENTS:
Time Frame: The AE reporting period was from consent until the subject's final study visit (Week 52). In addition, any untoward event that may occur subsequent to the reporting period that the Investigator assessed as possibly, probably or definitely related to the study drug medication was reported as an AE.
Arm/Group | Biktarvy | Symtuza
All-Cause Mortality (participants affected / at risk) | 9/220 | 3/222
Serious Adverse Events (participants affected / at risk) | 52/220 | 54/222
Other Adverse Events (participants affected / at risk) | 111/220 | 120/222
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Biktarvy (N=220) | Symtuza (N=222)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Acute appendicitis (Infections and infestations) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 2 (2)
Acute renal failure (Renal and urinary disorders) | 1 (2) | 1 (1)
Alcohol intoxication (Injury, poisoning and procedural complications) | 1 (1) | 1 (2)
Altered state of consciousness (Psychiatric disorders) | 0 (0) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Atypical mycobacterial pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Balance disorder (Nervous system disorders) | 0 (0) | 1 (1)
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Behavioural disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Bicytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Bilateral pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Breast ductal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 2 (2) | 0 (0)
Cardiac ischemia (Cardiac disorders) | 1 (1) | 0 (0)
Cellulitis of toe (Infections and infestations) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
Clostridium colitis (Infections and infestations) | 1 (1) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 1 (1)
Clostridium difficile infection (Infections and infestations) | 1 (1) | 1 (2)
Clostridium difficile sepsis (Infections and infestations) | 1 (1) | 0 (0)
CMV pneumonitis recurrent (Infections and infestations) | 0 (0) | 1 (1)
CMV retinitis (Infections and infestations) | 1 (1) | 0 (0)
CNS-IRIS (Nervous system disorders) | 0 (0) | 1 (2)
Cognitive impairment (Nervous system disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Community acquired pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Condyloma excision (Surgical and medical procedures) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1)
Cryptococcal meningitis (Infections and infestations) | 1 (1) | 0 (0)
Cytomegalovirus infection (Infections and infestations) | 2 (2) | 1 (1)
Cytomegalovirus infection reactivation (Infections and infestations) | 0 (0) | 1 (1)
Cytomegalovirus viraemia (Infections and infestations) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 2 (2)
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Diplopia (Eye disorders) | 0 (0) | 1 (1)
DRESS syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Drug eruption NOS (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Drug-induced hepatotoxicity (Hepatobiliary disorders) | 0 (0) | 1 (1)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Epiglottitis (Infections and infestations) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (5) | 0 (0)
Fever (General disorders) | 3 (3) | 3 (3)
Fever of unknown origin (General disorders) | 0 (0) | 2 (2)
Gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gonococcal arthritis (Infections and infestations) | 1 (1) | 0 (0)
Granulomatous disease (General disorders) | 0 (0) | 1 (1)
Haemophilus pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Hepatopathy (Hepatobiliary disorders) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 0 (0) | 2 (2)
HIV encephalopathy (Infections and infestations) | 0 (0) | 1 (1)
HIV with persistent generalized adenopathy (Infections and infestations) | 1 (1) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Immune reconstitution inflammatory syndrome (Immune system disorders) | 5 (5) | 1 (1)
Immune reconstitution syndrome (Immune system disorders) | 0 (0) | 1 (1)
Infection mycobacterium avium (Infections and infestations) | 1 (1) | 0 (0)
Intestinal pseudo-obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intra-abdominal abscess (Infections and infestations) | 0 (0) | 1 (1)
IRIS associated Kaposi's sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Kaposi sarcoma inflammatory cytokine syndrome (Infections and infestations) | 0 (0) | 1 (1)
Kaposi's sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Knee surgery NOS (Surgical and medical procedures) | 1 (1) | 0 (0)
Localised infection (Infections and infestations) | 1 (1) | 0 (0)
Loss of consciousness (Nervous system disorders) | 0 (0) | 1 (1)
Lymphocytic meningitis (Infections and infestations) | 0 (0) | 1 (1)
Malaise (General disorders) | 1 (1) | 0 (0)
Mastoiditis (Infections and infestations) | 0 (0) | 1 (1)
Mediastinal lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Mediastinal mass (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Methemoglobinemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Monkeypox (Infections and infestations) | 0 (0) | 1 (1)
Mycobacterial infection (Infections and infestations) | 1 (1) | 0 (0)
Mycobacterial infection NOS (Infections and infestations) | 1 (1) | 0 (0)
Mycobacterium avium complex immune restoration disease (Infections and infestations) | 0 (0) | 1 (1)
Mycobacterium avium complex infection (Infections and infestations) | 0 (0) | 1 (1)
Mycobacterium avium complex lymphadenitis (Infections and infestations) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Oesophageal candidiasis (Infections and infestations) | 0 (0) | 1 (1)
Opportunistic infection (Infections and infestations) | 1 (1) | 0 (0)
Pancolitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pelvic fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Pneumocystis jirovecii infection (Infections and infestations) | 1 (1) | 0 (0)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Pneumocystis pneumonia (Infections and infestations) | 2 (2) | 0 (0)
Pneumocystosis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 4 (4) | 2 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Polytrauma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Posterior uveitis (Infections and infestations) | 1 (1) | 0 (0)
Progressive multifocal leukoencephalopathy (Infections and infestations) | 0 (0) | 2 (2)
Pseudomonas infection (Infections and infestations) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pulmonary tuberculosis (Infections and infestations) | 1 (1) | 0 (0)
Purulent pericarditis (Infections and infestations) | 1 (1) | 0 (0)
Pustular rash (Infections and infestations) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Reiter syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Renal calculi (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rhinovirus infection (Infections and infestations) | 0 (0) | 1 (1)
Rhodococcus equi infection (Infections and infestations) | 1 (1) | 0 (0)
SARS-CoV-2 infection (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Septic arthritis (Infections and infestations) | 0 (0) | 1 (1)
Septic shock (Infections and infestations) | 2 (2) | 0 (0)
Skin rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Stereotactic needle biopsy of breast (Investigations) | 0 (0) | 1 (1)
Stomach flu (Infections and infestations) | 0 (0) | 1 (1)
Swelling (r) testicle (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Thrombosis leg (Vascular disorders) | 0 (0) | 1 (1)
Toxoplasmosis recurrent (Infections and infestations) | 0 (0) | 1 (1)
Transcervical fracture, open (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Traumatic shock (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tuberculosis (Infections and infestations) | 0 (0) | 2 (2)
Upper gastrointestinal bleeding (Gastrointestinal disorders) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1)
Viral pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Visual acuity lost (Eye disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0)
Respiratory infection (Infections and infestations) | 1 (1) | 0 (0)
Alcohol intoxication acute (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Drug Overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Drug rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Biktarvy (N=220) | Symtuza (N=222)
Cough (Respiratory, thoracic and mediastinal disorders) | 15 (16) | 16 (16)
COVID-19 (Infections and infestations) | 13 (13) | 15 (15)
Diarrhea (Gastrointestinal disorders) | 13 (14) | 9 (11)
Diarrhoea (Gastrointestinal disorders) | 11 (11) | 17 (18)
Fever (General disorders) | 16 (20) | 12 (15)
Headache (Nervous system disorders) | 20 (23) | 22 (25)
Hypertension (Vascular disorders) | 16 (17) | 10 (10)
Insomnia (Psychiatric disorders) | 16 (16) | 15 (16)
Nausea (Gastrointestinal disorders) | 16 (16) | 21 (23)
Rash (Skin and subcutaneous tissue disorders) | 13 (13) | 17 (22)
Weight gain (Investigations) | 13 (13) | 10 (10)
Constipation (Gastrointestinal disorders) | 6 (7) | 14 (14)
Oral Candiasis (Infections and infestations) | 4 (5) | 15 (15)
Vitamin D deficiency (Metabolism and nutrition disorders) | 7 (7) | 12 (12)
Vomiting (Gastrointestinal disorders) | 5 (5) | 15 (15)

LIMITATIONS AND CAVEATS:
The open-label design may have influenced AE reporting, although objective outcomes were adjudicated The 48-week follow-up limits insight into long-term outcomes such as metabolic effects, weight gain, and virological durability.

Excluding patients with active tuberculosis or cryptococcal meningitis restricts applicability to high-risk subgroups.

The predominantly European cohort may not reflect PWAD in regions with higher burdens of opportunistic infections.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-03-11): https://cdn.clinicaltrials.gov/large-docs/60/NCT03696160/Prot_SAP_000.pdf